CLINICAL TRIAL: NCT02361437
Title: Safety and Efficacy of Vasculera® in the Healing of Diabetic Skin Ulcers and Improving Insulin Sensitivity: A Pilot Study
Brief Title: Safety and Efficacy of Vasculera® in the Healing of Diabetic Skin Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator's hospital sold and study cancelled without enrollment.
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PVD-01
Record Dates: First submitted 2015-02-04; First posted 2015-02-11 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2015-10

CONDITIONS: Diabetic Ulcers
Keywords: diabetes type II; diabetic ulcers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diosmin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Vasculera
- Vasculera (Experimental): diosmin
  Interventions: Dietary Supplement: Vasculera

INTERVENTIONS:
Dietary Supplement: Vasculera — Vasculera 630 mg b.i.d.
  Other Names: diosmin

SUMMARY:
This study is designed to evaluate if Vasculera, a marketed medical food product, will improve the rate and extent of healing of diabetic ulcers.

DETAILED DESCRIPTION:
This study is designed primarily to compare the rate and extent of healing of diabetic ulcers in people treated with or without Vasculera while maintaining a standard of care (SOC) therapeutic regimen. The study will also examine the effects of Vasculera on anti-diabetic medication requirements and markers of microvascular disease. Subjects will be stratified by whether or not they receive hyperbaric oxygen therapy (HBOT) as part of their SOC treatment regimen. In addition, the study will examine the ability of Vasculera to improve glycemic control and reduce anti-diabetic medication requirements (oral or injectable insulin) and will gather preliminary information on the ability of Vasculera to improve microvascular blood flow and oxygen delivery peripheral tissues including ulcerative lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender, between 25-85 years old
2. Diagnosis of type II diabetes
3. Presence of a grade I-III skin ulcer of diabetic origin and at least 1 cm in diameter for more than 60 days and not improving despite standard conventional care without HBOT
4. Treatment with oral anti-diabetic agents and/or insulin for at least 1 year. Dose must be stable for at least 3 months.
5. Not using any other product for control of serum glucose including medical foods, neutraceuticals or dietary supplements
6. Consistent dietary habits
7. Able to understand and sign informed consent document

Exclusion Criteria:

1. age less than 25 years or greater than 85 years
2. Skin ulceration of other than diabetic etiology
3. diagnosis of type I diabetes
4. use of any other serum glucose modifying agent, other than stable prescribed anti-diabetic medication regimen within 12 weeks of screening visit
5. use of nutritional supplements specifically for anti-oxidative purposes (e.g., multivitamins allowed)
6. history of collagen vascular disease
7. taking corticosteroids in any dose, by any route
8. no history of therapy with pentoxyphylline or cilostazol for 2 months prior to the screening visit and for the duration of the study
9. history of any intestinal disease that might interfere with absorption of study products
10. any active malignancy or history of malignancy within 3 years of the screening visit,, except basal cell carcinoma or cervical carcinoma in situ curatively treated
11. screening AST, ALT, alkaline phosphatase, bilirubin >1.3 times the upper limit of normal for the reference laboratory
12. serum creatinine >3.0
13. diabetes mellitus not on stable therapy for at least 3 months
14. history of chronic pancreatitis
15. uncontrolled hypertension (DBP >100, SPB >160)
16. unstable angina, other uncontrolled cardiac disease including NYHA CHF Class III or IV
17. pregnant or lactating women
18. known history of allergies to citrus, diosmin, or Alka-4 Complex
19. history of substance abuse, or any psychiatric condition that may impair the subject's ability to comply with the study requirements.
20. Consumption of more than one (1) unit of alcohol daily. For the purposes of this study a unit of alcohol is defined as 12 oz. of beer, 6 oz. of wine or 1.5 oz. of hard spirits
21. Concomitant use of chlorzoxazone, diclofenac or metronidazole
22. any medical condition that, in the opinion of the investigator, might put the subject at undue risk or might interfere with the subject's ability to participate in the study
23. participation in another clinical trial within 30 days or 7 half-lives of the prior study product, whichever is longer, of the screening visit

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of healing of diabetic ulcers measured by ulcer size | 4 months
  days to complete healinh

SECONDARY OUTCOMES:
Efficacy of diabetic control measure by reduction of oral anti-diabetic medication and/or insulin requirements | 4 months
  anti-diabetic medication doses
Reduction on peripheral edema measured by leg circumferance | 4 months
  leg circumference
lower extremity skin oxygenation measured by trancutaneous oximetry | 4 months
  transcutaneous oximetry at toes

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Levy, MD, Study Director — Primus Pharmaceuticals, Inc
Locations (1):
- Nix Hospital, San Antonio, Texas, United States